CLINICAL TRIAL: NCT05362136
Title: Assessment of the Effect of Sinus Floor Perforation During Sinus Floor Elevation on Bone Formation Within the Augmentation Material
Brief Title: Effect of Multiple Perforations of the Sinus Floor on Bone Formation After Sinus Floor Elevation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Kristina Bertl, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1709/2016
Record Dates: First submitted 2022-05-01; First posted 2022-05-05 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Sinus Elevation; Dental Implant; Bone Formation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): standard sinus floor elevation
  Interventions: Procedure: no perforation of the sinus floor
- Test (Experimental): standard sinus floor elevation with additional perforation of the sinus floor
  Interventions: Procedure: perforation of the sinus floor

INTERVENTIONS:
Procedure: perforation of the sinus floor — perforation of the cortical layer of the sinus floor prior to inserting the augmentation material during sinus floor elevation
  Arms: Test
Procedure: no perforation of the sinus floor — standard procedure for sinus floor elevation
  Arms: Control

SUMMARY:
The aim of the present study is to compare the rate of new bone formation after sinus floor elevation with or without perforation of the cortical sinus floor prior to insertion of augmentation material. Twelve patients requiring bilateral sinus floor elevation will be recruited for a pilot study in split-mouth design. On both sides a lateral window will be prepared and the sinus mucosa will be elevated. After this step, the sides are assigned as test or control side. While the control side is just filled with augmentation material, an additional step is performed for the test side, i.e., prior to inserting the augmentation material, the cortical bone layer of the sinus floor is perforated several times into the trabecular bone layer to improve the blood supply to the grafting material. Thereafter, both sides are left to healing for 4-6 months until implant installation. At timepoint of implant installation, a bone biopsy will be collected to allow histological assessment of the grafted area.

ELIGIBILITY:
Inclusion Criteria:

* in need of bilateral sinus floor elevation
* residual alveolar ridge height 2-6mm
* residual alveolar ridge width > 4mm

Exclusion Criteria:

* uncontrolled periodontal disease
* acute or chronic sinusitis

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-03-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
New bone formation | 4-6 months after sinus floor elevation
  histological assessment of new bone formation after sinus floor elevation (%)

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Dentistry, Medical University of Vienna, Vienna, Austria